CLINICAL TRIAL: NCT05079841
Title: The Stimulation To Induce Mothers (STIM) Study: A Parallel Group Randomized Controlled Trial
Brief Title: The Stimulation To Induce Mothers Study
Acronym: STIM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000031338; 1R01HD111633-01 (NIH); 231888-1 (Other Grant/Funding Number: Cornell University, Joan and Sanford I. Weill Medical College)
Record Dates: First submitted 2021-09-20; First posted 2021-10-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Oxytocin; Labor Pain; Induction of Labor Affected Fetus / Newborn; Physiologic Effects of Drugs
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intrapartum nipple stimulation (Experimental): Participants randomized to the intrapartum nipple stimulation will use electric breast pump or stimulate by hand (intervention) to induce labor.
  Interventions: Device: Electric breast pump
- Exogenous oxytocin intravenous infusion (Active Comparator): Participants randomized to the standard care arm will use exogenous oxytocin intravenous infusion to induce labor.
  Interventions: Drug: Exogenous oxytocin intravenous infusion without nipple stimulation.

INTERVENTIONS:
Device: Electric breast pump — Participants randomized to the intrapartum nipple stimulation will use electric breast pump or nipple stimulate by hand (if preferred) (intervention) to induce labor for at least 2 hours
  Arms: Intrapartum nipple stimulation
Drug: Exogenous oxytocin intravenous infusion without nipple stimulation. — Participants randomized to the standard care arm will use exogenous oxytocin intravenous infusion to induce labor as current standard of care
  Other Names: Pitocin intravenous infusion
  Arms: Exogenous oxytocin intravenous infusion

SUMMARY:
The investigators propose a parallel group randomized clinical trial of intrapartum nipple stimulation versus exogenous oxytocin infusion for nulliparous women undergoing induction of labor near term. The central hypothesis is that intrapartum nipple stimulation to induce labor increases spontaneous vaginal delivery, improves patient-centered outcomes such as childbirth satisfaction, labor agentry, and pain scores, and reduces adverse neonatal and maternal outcomes in nulliparous women. The investigators will pursue the following specific aims: 1) Assess the effectiveness of intrapartum nipple stimulation on the rate of spontaneous vaginal delivery in nulliparous women, 2) Breastfeeding as the sole source of nutrition at time of maternal hospital discharge (Primary Aims); 3) Maximal percent newborn weight loss during the birth hospitalization within 72 hours of life, 4) Determine the effect of intrapartum nipple stimulation on the rate of adverse maternal and neonatal outcomes, 5) Determine the impact of intrapartum nipple stimulation on patient-centered outcomes and 6) In a sub-cohort of women who are enrolled in the trial, investigators will measure the change in oxytocin concentration from baseline to time at which patient achieves a regular contraction pattern.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine whether intrapartum nipple stimulation therapy with or without synthetic oxytocin changes the likelihood of achieving a spontaneous vaginal delivery compared to receipt of synthetic oxytocin infusion without nipple stimulation to induce labor.
2. Breastfeeding as the sole source of nutrition at time of maternal hospital discharge

Secondary Objectives (if applicable)

The secondary objectives are as follows:

1. Determine whether intrapartum nipple stimulation therapy with or without synthetic oxytocin changes the likelihood of achieving a spontaneous vaginal delivery compared to receipt of synthetic oxytocin infusion without nipple stimulation to induce labor.
2. Determine if women who perform intrapartum nipple stimulation to induce labor have differences in other obstetric and maternal outcomes
3. Determine if women who perform intrapartum nipple stimulation report differences in pain scores during labor, labor agentry and satisfaction scores, postpartum depression scores, and breastfeeding success compared to women who receive only intrapartum exogenous oxytocin infusion.
4. Determine if women who perform intrapartum nipple stimulation to induce labor have similar fetal and neonatal outcomes compared to women who receive only intrapartum exogenous oxytocin infusion.
5. Maximal percent newborn weight loss during the birth hospitalization within 72 hours of life
6. At Yale, to measure the change in oxytocin concentration from baseline over the course of labor induction in patients undergoing induction of labor via intrapartum nipple stimulation versus continuous exogenous oxytocin infusion.
7. At Yale, to measure circulating plasma and urine concentrations of proteins, microRNA, and small molecules using unbiased "omics" approaches, comparing patients undergoing induction of labor via intrapartum nipple stimulation versus continuous exogenous oxytocin infusion, un-ripened/unlabored control patients, and patients in spontaneous labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Gestational age 36 0/7 weeks and greater at enrollment
* Singleton gestation
* Planned to undergo initiation of exogenous oxytocin infusion by their maternity care provider
* Spontaneous rupture of membranes or if membranes intact, modified Bishop score ≥5 and cervix dilated <6 cm within one hour of enrollment
* Ability to give informed consent

Exclusion Criteria:

* Unable to understand English or Spanish
* Prior use of exogenous oxytocin or attempt at nipple stimulation during the current pregnancy
* Presence of tachysystole (defined as more than 5 contractions in 10 minutes averaged over 30 minutes), recurrent variable or late fetal decelerations, and bradycardia in the prior 30 minutes before enrollment
* Non-vertex presenting fetus at time of enrollment
* Planned for cesarean delivery or contraindication to labor by institutional policy (e.g., placenta previa, vasa previa, active genital herpes infection, previous transmural myomectomy)
* Multi-fetal gestation (e.g., twins, triplets, and higher-order multiples)
* Intrauterine fetal death
* Major fetal anomaly suspected prenatally (defined as a fetal anomaly with anticipated neonatal intensive care unit admission)
* Suspected alloimmunization (given the increased likelihood for anticipated neonatal intensive care unit admission)
* Known severe fetal growth restriction (estimated fetal weight <3rd percentile) or abnormal umbilical artery Doppler studies (given the increased likelihood for anticipated neonatal intensive care unit admission)
* HIV infection (nipple stimulation is not encouraged given the recommendation for these mothers not to breastfeed)
* Participation in another interventional study that influences management of labor and delivery or perinatal morbidity or mortality
* History of mastectomy or other contraindication to use of electronic breast pump
* Known allergic reactions to components of the electronic breast pump or to synthetic oxytocin intravenous solution
* Significantly impaired consciousness or executive function (e.g., intubated or sedated)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 988 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Spontaneous vaginal delivery | At delivery
  Spontaneous vaginal delivery will be defined as delivery that occurs without the use of forceps, vacuum, or cesarean
Breastfeeding as the sole source of nutrition (BSSN) | up to 72 hours following delivery
  Number of participants using breastfeeding as the sole source of nutrition (BSSN) at time of maternal discharge or 72 hours of life (whichever is sooner)

SECONDARY OUTCOMES:
Operative vaginal delivery | At delivery
  Delivery with the assistance of forceps or vacuum, and indication
Cesarean delivery | At delivery
  Delivery by cesarean section
Labor induction duration | At delivery
  Time interval from randomization to delivery
Number of Participants with Postpartum hemorrhage | From delivery to 24 hours postpartum
  Cumulative blood loss of ≥1,000 mL within 24 hours after the birth process
Number of Participants with Severe Postpartum hemorrhage | From delivery to 24 hours postpartum
  Transfusion; non-elective hysterectomy; use of ≥2 uterotonic medications other than oxytocin; other interventions such as uterine compression sutures, uterine artery ligation or embolization, hypogastric artery ligation, balloon tamponade
Number of participants with suspected infection | 3-7 days postpartum
  Suspected intraamniotic infection, intrapartum chorioamnionitis, or postpartum endometritis (defined as maternal fever ≥38° Fahrenheit with planned or initiated administration of therapeutic antibiotics) after randomization and prior to delivery hospitalization discharge
Lactational mastitis | After delivery to 12 weeks postpartum
  Subject-reported occurrence of lactational mastitis
Number of maternal deaths | immediately prior to up to immediately post delivery
  Incidence of maternal death prior to, during, or post delivery
Maternal Intensive Care Unit admission | 3-7 days postpartum
  Any admission to the Intensive Care Unit after delivery and prior to delivery hospitalization discharge
Neonatal Intensive Care Unit admission | up to 28 days following birth
  Any admission to the Neonatal Intensive Care Unit From birth to birth hospitalization discharge or 28 days after birth, whichever is earlier
Neonatal Apgar score ≤3 at 5 minutes of life | At 5 minutes after birth
  The Neonatal Apgar score is scored from 0 to 10. A 5-minute Apgar score of 0-3 correlates with neonatal mortality in large population studies.
Umbilical acidemia | At delivery
  Umbilical cord arterial pH <7.0 or base excess >12 mmol/L; or umbilical cord venous pH <7.0 or base excess >12 mmol/L if arterial blood sample not available
Composite neonatal severe morbidity measure | up to 28 days following delivery
  Intrapartum fetal death or neonatal death; cardiorespiratory support within first 72 hours of life; neonatal encephalopathy; seizures; hypothermic treatment (cooling); sepsis; pneumonia; major birth injury; meconium aspiration syndrome; intracranial hemorrhage or subgaleal hemorrhage; or hypotension requiring pressor support
Percent newborn weight loss | At 72 hours of life or birth hospitalization discharge, whichever is earlier
  Maximal percent newborn weight loss in kilograms(kg)

OTHER OUTCOMES:
Subject-reported pain during childbirth | At intervention start and than again 2 hours after intervention start
  Visual analog scale, scored with Likert scale from 0 (no pain) to 10 (worst pain)
Subject-reported satisfaction during labor and childbirth | 6-96 hours after delivery
  Birth Satisfaction Scale-Revised (BSS-R) is a 10-item self-report valid and reliable measure (scores range from 0 to 40, 0 being the least satisfaction and 40 being the most satisfaction)
Subject-reported feelings of control during labor and childbirth | 6-96 hours after delivery
  Labor Agentry Scale is a 29-item survey designed to assess expectations and experiences of personal control during childbirth (scores range from 29 to 203, with higher scores indicating greater perceived control during childbirth)
Subject-reported depression score | 4 to 12 weeks after delivery
  Edinburgh Postnatal Depression Scale is a 10-item self report scored from 0 to 30; score >10 warrants additional clinical assessment for depression
Subject-reported breastfeeding success | 4 to 12 weeks after delivery
  Maternal Breastfeeding Evaluation Scale (MBES) is a 30-item using a 5-point Likert scale with higher scores reflecting more positive breastfeeding experiences.
Subject-reported ability to express and/or collect colostrum and/or breastmilk intrapartum | From randomization to hospital discharge, approximately 3-7 days
  Participants ability to express and/or collect colostrum and/or breastmilk intrapartum
Subject-reported perception of milk supply | 2 weeks postpartum
  Subject-reported perception of milk supply using the validated Perception of Insufficient Milk Supply (PIMS). PIM is defined as a state in which a mother has or perceives that she has an inadequate supply of breast milk to meet her infant's needs. A perception of insufficient milk supply is associated with early discontinuation of breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Molly McAdow, MD, PhD, Principal Investigator — Yale University; Bethany Stetson, MD, Principal Investigator — Northwestern University; Moeun Son, MD, MSCI, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with academic researchers for secondary analyses or meta-analyses only after approval from the principal investigator and using an IRB-approved mechanism.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available after publication and will be available for 5 years.
Access Criteria: De-identified data will be shared with academic researchers for secondary analyses or meta-analyses only after approval from the principal investigator and using an IRB-approved mechanism.

REFERENCES:
- [Derived] Tortal D, Shabanova V, Taylor S, Xu X, McAdow M, Stetson B, McCollum S, Sanchez E, Adjakple A, Leventhal J, Son M. Stimulation Therapy to Induce Mothers: Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2024 Aug 29;13:e63463. doi: 10.2196/63463. PMID 39207839

DOCUMENTS (2):
  • Study Protocol (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT05079841/Prot_001.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT05079841/ICF_000.pdf